CLINICAL TRIAL: NCT03978065
Title: The Renal Transplant Outcome Prediction and Validation Study (TOPVAS)
Brief Title: The Renal Transplant Outcome Prediction and Validation Study
Acronym: TOPVAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Version 1.1
Record Dates: First submitted 2019-03-04; First posted 2019-06-06 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-03

CONDITIONS: Ischemia Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Microscopy, Confocal

STUDY DESIGN:
Intervention Model Description: Prospective, single-center pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Confocal microscopy — For this purpose "live stains" will be combined with a confocal imaging setup equipped with 6 laser lines. A major advantage of this technique is that tissue specimens do not need to be fixed prior to analysis. Such an approach does not only allow tissue viability and integrity assessment in an unprecedented speed and accuracy, but also promises to shed new light into quality assessment and prognosis in kidney transplantation. The investigators herein wish to establish the predictive values of this technology in kidney transplantation.
  The methodology used in this trial is referred to as BIOPSYCHRONOLOGY - as a reference to dendrochronology, or tree ring dating. Leaving the biopsy sample intact facilitates its analysis, just as drills are used for tree-ring counting.

SUMMARY:
The number of patients with end stage renal disease is increasing continuously and kidney transplantation is the preferred treatment modality. Modern immunosuppressive therapy has reduced the number of acute rejection episodes and increased one year allograft survival dramatically. Nonetheless, 4% of allografts are lost beyond the first year annually due to a multifactorial process and the latter number has not changed for decades. One of the most important factors to determine long-term success after kidney transplantation is the quality of the donor organ. For example, transplantation of organs from elderly or extended criteria donors results in reduced allograft and patient survival.

In previous work, the investigators specifically focused on age-associated molecular signatures including telomere length and mRNA expression levels of the cell cycle inhibitors CDKN2A (p16INK4a) and CDKN1A (p21WAF1) and assessed these parameters in pre-implantation biopsies of 54 patients. In a linear regression analysis CDKN2A turned out to be the best single predictor for serum creatinine after 1 year followed by donor age and telomere length. A multiple linear regression analysis revealed that the combination of CDKN2A values and donor age yielded even higher predictive values. In another study the investigators were able to show an interaction between donor age and use of calcineurin inhibitors with regard to outcome after renal transplantation.

During these past activities an extensive set of whole genome transcriptomics profile information from zero hour biopsies and clinical follow-up data has been collected. In the TOPVAS study, existing data derived from 72 of the above mentioned set of biopsies (exclusion of live donor grafts) will be analysed with state of the art bioinformatical/system biology tools to derive a general (not purely age associated) prognostic biomarker panel for functional transplant outcome two years after transplantation. This marker panel will also be used to define organs preferentially suitable for MMF/tacrolimus based immunosuppression. Both panels will then be validated for their prognostic and predictive information on the long-term outcome after transplantation in a new independent patient population treated with tacrolimus and MMF. In addition to biomarker assessment and in pursue of identifying alternative and/or complementary parameters with predictive value , an advanced morphological investigation of tissue biopsy life stains will be performed employing an innovative cell viability staining technology ("BIOPSYCHRONOLOGY").

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Recipient age > 18 years
* First or second deceased donor kidney transplantation
* Panel reactive antibody frequency <50%

Exclusion Criteria:

* Combined kidney transplantation with another organ
* Living donor kidney transplantation
* TOPVAS is a interventional prospective cohort study and participation of patients in other randomized prospective interventional trials does not per se violate the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
The number of dialysis in the first 7 days post transplant | 7 days
  The need of at least one dialysis within the first 7 days post transplant.
Kidney parenchyma quality | before transplant
  Live and dead cells in the kidney biopsy will be quantified using the dyes Syto-16/PI and WGA will be calculated as follows:
  Groups: The number of dead/live cells will be entered in the following groups
  1. Total count (irrespective of localization).
  2. Tubular area (cells from the tubular area)
  3. Glomerular area (cells from the glomerulus) For each group the number of viable cells will be divided by the number of dead cells.
  (+1) Using this approach we will obtain for highly viable biopsies/areas high numbers, bigger than (0) For biopsies/areas in which the number of viable cells equals the one of dead cells we will obtain 1.
  (-1) For those in which the number of dead cells outnumbers the one of live cells, numbers between 1 and 0 will be obtained.
  For each biopsy, a score will be calculated which will consist of the two tubular areas and the glomerular area. Therefore a maximum of +3 points can be achieved, or in the worst case -3.

IPD SHARING:
Plan to Share IPD: No